CLINICAL TRIAL: NCT03923751
Title: Survey of Regional Anesthesia Practice in Poland - National Survey 2018
Brief Title: Survey of Regional Anesthesia Practice in Poland
Acronym: AnkietaRA
Status: Completed | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Collaborators: Department of Anesthesiology and Intensive Care, Czerniakowski Hospital, Warsaw (Unknown); Polskie Towarzystwo Znieczulenia Regionalnego i Leczenia Bólu (Polish ESRA) (Unknown); Sekcja Znieczulenia Regionalnego i Terapii Bólu, Polskie Towarzystwo Anestezjologii i Intensywnej Terapii (PTAiIT) (Unknown)
Responsible Party: Principal Investigator, Marek Janiak, Doctor, Medical University of Warsaw
Other Study IDs: Ankieta RA 2018
Record Dates: First submitted 2019-04-18; First posted 2019-04-23 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Anesthesia, Regional

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Polish Hospitals: Hospitals with anesthesia or intensive care practices
  Interventions: Other: Invitation to regional anesthesia survey

INTERVENTIONS:
Other: Invitation to regional anesthesia survey — An invitation letter sent to Head of Anesthesiology and Intensive Care Department of Polish Hospital

SUMMARY:
The study is being conducted to gain insight into regional anesthesia practice in polish hospitals specifically asking for methods used, accessibility to equipment and preference for regional blockade and perioperative analgesia.

DETAILED DESCRIPTION:
In recent years, regional anesthesia has become one of the most dynamic parts of anesthesiology. This is in part due to less invasive surgical procedures, surgical enhanced recovery protocols as well as the incorporation of ultrasonography into the daily practice of regional anesthesia.

The aim of this retrospective survey is to track and analyse the changes in everyday practice of regional anesthesia in Poland that have occurred in the year 2018.

An invitation to the survey will be sent to all heads of anesthesiology departments in Poland. The answers to the survey will be collected using an internet based website created by the authors of the study.

ELIGIBILITY:
Inclusion Criteria:

* All Polish hospitals practising anesthesiology and intensive care in the national register of medical practices (www.rpwdl.csioz.gov.pl)

Exclusion Criteria:

* Hospitals and medical practices not practising anesthesiology or intensive care

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Anesthetists in Polish Hospitals
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Regional anesthesia practice | Up to 12 months practice in the year 2018
  Answers of head of anesthesiology and intensive care departments regarding regional anesthesia practice in their respective department by completing the Regional Anesthesia Survey 2018: multiple and single choice answers
Regional anesthesia practitioners | Up to 12 months in the year 2018
  Answers of head of anesthesiology and intensive care departments regarding number of anesthesiologists practicing regional anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- I Department of Anesthesiology and Intensive Care Warsaw Medical University, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No
Results will be published only as collective data